CLINICAL TRIAL: NCT01908699
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled, Phase 3 Study to Assess the Efficacy and Safety of Oral BPS-314d-MR added-on to Treprostinil, Inhaled (Tyvaso®) in Subjects With Pulmonary Arterial Hypertension
Brief Title: Beraprost-314d Added-on to Tyvaso® (BEAT)
Acronym: BEAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lung Biotechnology PBC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BPS-314d-MR-PAH-302
Record Dates: First submitted 2013-07-16; First posted 2013-07-26 (Estimated); Results first posted 2020-02-28 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — beraprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Beraprost Sodium 314d Modified Release Tablets (Experimental): Available as 15 μg tablets for oral, 1 or 2 tablets four times daily (QID) administration.
  Interventions: Drug: Beraprost Sodium 314d Modified Release Tablets
- Placebo (Experimental): Placebo tablets, which are identical in size and appearance to those containing BPS-314d-MR.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Beraprost Sodium 314d Modified Release Tablets — Available as 15 μg tablets for oral, 1 or 2 tablets four times daily (QID) administration
  Arms: Beraprost Sodium 314d Modified Release Tablets
Drug: Placebo — Placebo tablets, which are identical in size and appearance to those containing BPS-314d-MR
  Arms: Placebo

SUMMARY:
This is a multicenter, double-blind, randomized, placebo-controlled Phase 3 study, to assess the efficacy and safety of BPS-314d-MR when added-on to inhaled treprostinil (Tyvaso®)in patients with pulmonary arterial hypertension.

Patients new to Tyvaso, will enter a run-in period on inhaled treprostinil until 90 days of experience is achieved to ensure drug tolerability before enrolling in the study.

Treatment groups consist of one active and one placebo group. Subjects will be randomly allocated in a 1:1 ratio to one of the two treatment groups.

ELIGIBILITY:
Inclusion Criteria

The following are inclusion criteria to be enrolled in this study:

1. Male or female, age 18 to 80 years (inclusive).
2. Established diagnosis of pulmonary arterial hypertension that is either idiopathic or familial PAH, collagen vascular disease associated PAH, PAH associated with HIV infection, PAH induced by anorexigens/toxins, or PAH associated with repaired congenital systemic-to-pulmonary shunts (repaired ≥1 years).
3. If HIV positive, has a CD4 lymphocyte count ≥200 cells/mm3 within 30 days of Baseline Visit and is receiving current standard of care antiretroviral or other effective medication.
4. At the Screening Visit, WHO functional class III or IV and who have declining or unsatisfactory clinical response to current PAH therapy.
5. At the Baseline Visit, WHO functional class III or IV and who have declining or unsatisfactory clinical response to inhaled treprostinil therapy.
6. Able to walk unassisted (oxygen use allowed).
7. A 6-Minute Walk distance (6MWD) of ≥ 100 meters at the Screening Visit.
8. Previous (within five years prior to the Baseline Visit) right heart cardiac catheterization (RHC) with findings consistent with PAH, specifically mean Pulmonary Arterial Pressure (PAPm) ≥25 mmHg (at rest), Pulmonary Capillary Wedge Pressure (PCWP) (or left ventricular end diastolic pressure) ≤15 mmHg, and Pulmonary Vascular Resistance (PVR) >3 mmHg/L/min.
9. Echocardiography excluding any clinically significant left heart disease (e.g. left sided valve disease, wall motion abnormality suggesting of myocardial infarction, left ventricular hypertrophy, etc).
10. Pulmonary function tests conducted within 12 months before or during the Screening period to confirm the following:

    1. Total lung capacity (TLC) is at least 60% (predicted value) and
    2. Forced expiratory volume at one second (FEV1) of at least 50% (predicted value).
11. Subjects receiving additional FDA approved PAH therapies must be stable on their current dose for at least 30 days prior to the Baseline Visit, apart from modification of anticoagulant or diuretic dosages.
12. Must have completed 90 days of uninterrupted inhaled treprostinil treatment and received a stable dose of inhaled treprostinil for at least 30 days prior to Baseline to be eligible for randomization into the study.
13. Women of child-bearing potential (defined as less than 1 year post-menopausal and not surgically sterile) must be practicing abstinence or using two highly effective methods of contraception (defined as a method of birth control that result in a low failure rate, i.e., less than 1% per year, such as approved hormonal contraceptives, barrier methods [such as a condom or diaphragm] used with a spermicide, or an intrauterine device). Subject must have a negative pregnancy test at the Screening and Baseline Visits.
14. Willing and able to comply with study requirements and restrictions.

Exclusion Criteria

Patients who meet any of the following criteria will be excluded from the study:

1. Pregnant or lactating.
2. Has previous experience with beraprost or BPS-314d (i.e., BPS-IR, BPS-MR or BPS-314d- MR).
3. PAH related to any condition not covered under inclusion criteria, including but not limited to pulmonary venous hypertension, pulmonary veno-occlusive disease, pulmonary capillary hemangiomatosis, or chronic thromboembolic pulmonary hypertension.
4. History of interstitial lung disease, unless subject has collagen vascular disease and has had pulmonary function testing conducted within 12 months of the Baseline Visit demonstrating a total lung capacity ≥60% of predicted.
5. Has active hemorrhagic condition (e.g., upper digestive tract hemorrhage, hemoptysis, etc), or has a pre-existing condition that, in the Investigator's judgment, may increase the risk for developing hemorrhage during the study (e.g., hemophilia). Transient hemorrhage (e.g., epistaxis, normal menstrual bleeding, gingival bleeding, hemorrhoidal bleeding, etc) will not preclude enrollment.
6. Has received any investigational drug, device or therapy within 30 days prior to the Baseline Visit or is scheduled to receive another investigational drug, device or therapy during the course of the study.
7. Has any musculoskeletal disease or any other disease that would significantly limit ambulation.
8. Has any form of unrepaired or recently repaired (< 1 year) congenital systemic-to-pulmonary shunt other than patent foramen ovale.
9. Evidence of significant coronary arterial disease with symptoms, such as angina.
10. Left sided myocardial disease as evidenced by left ventricular ejection fraction < 40%, or shortening fraction <22%.
11. Has creatinine clearance <30 (using the Cockroft-Gault formula) or requires hemodialysis.
12. Has Childs-Pugh class C liver cirrhosis.
13. Has had previous atrial septostomy.
14. Any other clinically significant illness or abnormal laboratory values (measured during the Screening period) that, in the opinion of the Investigator, might put the subject at risk of harm during the study or might adversely affect the interpretation of the study data.
15. Anticipated survival less than 1 year due to concomitant disease.

The Sponsor recognizes that the pulmonary hypertension population is complex and diverse. In order to facilitate enrollment of appropriate subjects to this pivotal trial, Investigators are strongly encouraged to contact the medical director or study team to discuss potential study subjects who have comorbid conditions before enrollment into this study. See Appendix 9 for additional details.

No waivers to entry criteria are allowable in this study. Subjects who are initially ineligible for this study may be reassessed for eligibility after consultation with the Sponsor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2013-05-31 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-02-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (75):
- United States (69):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars-Sinai Medical Center Heart Institute, Beverly Hills, California
  - Allianz Research Institute Inc., Fountain Valley, California
  - University of California San Francisco - Fresno, Fresno, California
  - University of California - San Diego, La Jolla, California
  - University of California Los Angeles, Los Angeles, California
  - Keck Medical Center of USC, Los Angeles, California
  - Veterans Affairs Greater Los Angeles Healthcare System, Los Angeles, California
  - Center for Advanced Pulmonary Medicine, Rancho Mirage, California
  - University of California - San Francisco, San Francisco, California
  - Cottage Pulmonary Hypertension Center, Santa Barbara, California
  - Stanford University, Stanford, California
  - Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado Denver, Aurora, Colorado
  - Aurora Denver Cardiology Associates, Denver, Colorado
  - South Denver Cardiology Associates P.C., Littleton, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Bay Area Cardiology Associates, P.A., Brandon, Florida
  - Florida Lung, Asthma, and Sleep Institute, Celebration, Florida
  - University of Florida, Gainesville, Florida
  - University of Florida College of Medicine, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Florida Hospital, Orlando, Florida
  - Orlando Health Heart Institute, Orlando, Florida
  - South Miami Heart Specialists, South Miami, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Emory University, Atlanta, Georgia
  - Pulmonary & Critical Care of Atlanta, Atlanta, Georgia
  - Georgia Clinical Research, Austell, Georgia
  - Gwinnett Biomedical Research, Lawrenceville, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago Medicine, Chicago, Illinois
  - Advocate Health and Hospitals Corporation, Oakbrook Terrace, Illinois
  - Indiana University - Health Physicians, Carmel, Indiana
  - University of Iowa, Iowa City, Iowa
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - University of Louisville Department of Medicine, Louisville, Kentucky
  - John Ochsner Heart & Vascular Institute, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beaumont Health Systems, Troy, Michigan
  - Rutgers University Hospital, Newark, New Jersey
  - Albany Medical College, Albany, New York
  - Winthrop University Hospital, Mineola, New York
  - Beth Israel Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Pulmonary Health Physicians, PC, Syracuse, New York
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Anderson Pharmaceutical Research, Anderson, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Methodist Healthcare Clinical Trials Office, San Antonio, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Israel (6):
  - Soroka Medical Center, Beersheba
  - The Lady Davis Carmel Medical Center, Haifa
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 273 participants randomized, 271 received treatment: 136 participants in the esuberaprost group and 135 in the placebo group. Two participants were excluded after randomization and never received treatment: 1 participant in the esuberaprost group was randomized by mistake and 1 participant in the placebo group was terminated per physician decision.
Groups:
- Esuberaprost: Participants received 1 tablet of esuberaprost (BPS-314d-MR) 14.2 micrograms (mcg) orally 4 times daily (QID) (total daily dose: 56.8 mcg) in conjunction with inhaled treprostinil for 2 weeks. After 2 weeks, esuberaprost dose was increased to 2 tablets (14.2 mcg each) QID (total daily dose: 113.6 mcg). Participants who were unable to tolerate the 2 tablets QID dosing regimen were permitted to continue on 1 tablet QID during the study treatment.
- Placebo: Participants received 1 or 2 tablets of placebo matched to esuberaprost orally QID in conjunction with inhaled treprostinil.
Period: Overall Study
Arm/Group | Esuberaprost | Placebo
Started (Started = Randomized) | 137 | 136
Received at Least 1 Dose of Study Drug | 136 | 135
Completed | 62 | 58
Not Completed | 75 | 78
Not completed — Adverse Event | 8 | 12
Not completed — Lack of Efficacy | 2 | 2
Not completed — Lost to Follow-up | 2 | 4
Not completed — Physician Decision | 8 | 8
Not completed — Withdrawal by Subject | 15 | 10
Not completed — Pregnancy | 0 | 1
Not completed — Randomized in Error | 1 | 0
Not completed — Death | 9 | 12
Not completed — Progressive Disease | 30 | 29

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were collected on all randomized participants that received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Esuberaprost | Placebo | Total
Number analyzed (Participants) | 136 | 135 | 271
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.9 (13.61) | 56.1 (13.32) | 55.5 (13.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 98 | 197
  Male | 37 | 37 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 12 | 27
  Not Hispanic or Latino | 121 | 123 | 244
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 19 | 33
  White | 115 | 112 | 227
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 1 | 3
N-Terminal ProB-type Natriuretic Peptide (BNP) Levels [Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)] — BNP and NT-pro-BNP were used to detect, diagnose, and evaluate the severity of heart failure. Population: all randomized participants that received at least one dose of study drug and were analyzed for this baseline measure
  picograms per milliliter (pg/mL)
    number analyzed (Participants) | 113 | 105 | 218
    (all) | 99.65 (137.95) | 102.31 (240.51) | 100.93 (193.77)
Participant's Clinical Status Per World Health Organization (WHO) Functional Class [Count of Participants; unit: Participants] — Participant's clinical status was recorded according to the WHO functional class. Class I: No limitation of physical activities; Class II: Slight limitation of physical activities; Class III: Marked limitation of physical activities; and Class IV: Inability to carry out physical activities.
  Participants
    WHO Class I | 0 | 0 | 0
    WHO Class II | 0 | 0 | 0
    WHO Class III | 130 | 128 | 258
    WHO Class IV | 6 | 7 | 13
Borg Dyspnea Score [Mean (Standard Deviation); unit: score on a scale] — The Borg Dyspnea Scale is an 11-point scale used to rate the maximum level of dyspnea experienced during the 6MWT. Scores range from 0 (best condition) to 10 (worst condition) with nonlinear spacing of verbal descriptors of severity corresponding to specific numbers. At each scheduled study visit, subjects provided a rating of their dyspnea immediately following their 6MWT. Subjects could choose either the number or the verbal descriptor to reflect symptom intensity. Population: all randomized participants that received at least one dose of study drug and were analyzed for this baseline measure. 2. *In the case of a single, missing Baseline Day 1 or Day 2 Borg Dyspnea Score, the single value is used as Baseline Average value.
  score on a scale | 3.57 (1.91) | 3.84 (2.10) | 3.70 (2.01)
Six-Minute Walk Distance [Mean (Standard Deviation); unit: meters] — A 6 minute walk test (6MWT) was conducted that measured how far a participant could walk in 6 continous minutes. Participants were instructed to walk as far as possible in 6 minutes, and were allowed to slow down and take breaks as needed due to symptoms. Population: all randomized participants that received at least one dose of study drug and were analyzed for this baseline measure
  meters | 356.75 (109.32) | 365.37 (102.22) | 361.12 (105.62)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Experienced Clinical Worsening
Description: The number of participants that experienced a Clinical Worsening event confirmed by Endpoint Adjudication Committee at First Maximum Severity. Clinical Worsening was defined as any of these events following the Baseline visit: Death (all causes); Hospitalization due to worsening PAH; Initiation of a parenteral (infusion or sub-cutaneous) prostacyclin, directly related to worsening PAH; Disease progression; Unsatisfactory long-term clinical response.
  The number of participants that experienced clinical worsening is presented; time to clinical worsening data was not measured. Given the rate of clinical worsening overall and the large number of censored observations at the end of the study, the mean survival time estimates were not available for this endpoint.
Time Frame: up to 144 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Esuberaprost | Placebo
Number analyzed (Participants) | 136 | 135
Participants
  Death (all causes) | 8 | 13
  Hospitalization due to worsening PAH | 23 | 14
  Initiation of a parenteral prostacyclin | 7 | 13
  Disease progression | 6 | 4
  Unsatisfactory long-term clinical response | 5 | 7

2. Secondary Outcome: Mean Change From Baseline in Borg Dyspnea Score at Week 24
Description: The Borg dyspnea score was assessed prior to and following the completion of the 6MWT at Week 24. The Borg dyspnea score is a 10-point scale rating the maximum level of dyspnea experienced during the 6MWT. Scores range from 0 (for the best condition) to 10 (for the worst condition).
Time Frame: Baseline and Week 24
Population: Only participants with both a measurement at baseline and at the given visit are presented.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Esuberaprost | Placebo
Number analyzed (Participants) | 136 | 135
scores on a scale | -0.10 (1.68) | -0.26 (1.66)

3. Secondary Outcome: Mean Change From Baseline in NT-pro-BNP Levels at Week 24
Description: Plasma NT-proBNP concentration is a useful biomarker for PAH as it is associated with changes in right heart morphology and function.
Time Frame: Baseline and Week 24
Population: Only participants with both a measurement at baseline and at the given visit are presented.
Measure: Mean (Standard Deviation); unit: picomole per liter (pmol/L)
Arm/Group | Esuberaprost | Placebo
Number analyzed (Participants) | 136 | 135
picomole per liter (pmol/L) | 12.38 (131.46) | 20.48 (300.57)

4. Secondary Outcome: Change in WHO Functional Class From Baseline to Week 24
Description: Change from Baseline in participant clinical status was recorded according to the World Health Organization (WHO) Functional Class. A change from lower to higher functional class (i.e. 'III to IV' or 'II to III') was considered as a deterioration. A change from higher to lower functional class (i.e. 'III to II' or 'II to I') was considered as an improvement. All efficacy results are descriptive; no statistical analysis was conducted.
Time Frame: Baseline and Week 24
Population: Only participants with both a measurement at baseline and at the given visit are presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Esuberaprost | Placebo
Number analyzed (Participants) | 136 | 135
Participants
  Improved | 42 | 46
  No Change | 71 | 60
  Worsened | 0 | 2
  Not Reported | 23 | 27

5. Secondary Outcome: Mean Change From Baseline in Six Minutes Walk Distance (6MWD) at Week 24
Description: Area used for the Six Minute Walk Test (6MWT) was pre-measured at 30 meters in length. Rest periods were allowed if patient could no longer continue. If patient needed to rest, he/she could stand or sit and then begin again when rested but the clock continued to run. At the end of 6 minutes, the tester called "stop" while stopping the watch and then measured the distance walked. For purposes of the 6MWT, if patient was assessed at Baseline using oxygen therapy, all future 6MWT were conducted in the same manner.
Time Frame: Baseline and Week 24
Population: Only participants with both a measurement at baseline and at the given visit are presented.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Esuberaprost | Placebo
Number analyzed (Participants) | 109 | 106
meters | 13.47 (44.83) | 19.32 (53.23)

6. Secondary Outcome: Number of Participants With TEAEs, Serious TEAEs, Investigations SOC TEAEs, and Serious Investigations SOC TEAEs
Description: The number of participants experiencing overall Treatment-Emergent Adverse Adverse Events (TEAEs), serious TEAEs, Investigations SOC TEAEs, and serious Investigations SOC TEAEs were reported.Investigations SOC TEAEs were any event categorized within the Investigations System Order Class (SOC) and include adverse events due to physical examinations, vital signs, clinical laboratory parameters, and electrocardiogram findings.
Time Frame: up to 144 weeks
Population: Safety analysis population included all randomized participants who received at least 1 dose of study drug and analyzed as per the actual treatment received. Participants who received both esuberaprost and placebo were assigned to the esuberaprost group.
Measure: Number; unit: Participants
Arm/Group | Esuberaprost | Placebo
Number analyzed (Participants) | 137 | 134
Participants
  at least 1 TEAE | 135 | 132
  at least 1 Serious TEAEs | 75 | 78
  at least 1 Investigations SOC TEAEs | 61 | 49
  at least 1 Investigations SOC Serious TEAEs | 2 | 1

ADVERSE EVENTS:
Time Frame: Up to 144 weeks
Arm/Group | Esuberaprost | Placebo
All-Cause Mortality (participants affected / at risk) | 26/137 | 22/136
Serious Adverse Events (participants affected / at risk) | 75/137 | 78/136
Other Adverse Events (participants affected / at risk) | 135/137 | 132/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esuberaprost (N=137) | Placebo (N=136)
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Coagulopathy (Blood and lymphatic system disorders) | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 2 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 6
Atrial flutter (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 2 | 1
Cardiac failure (Cardiac disorders) | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 3
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Paroxysmal atrioventricular block (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 1
Pulseless electrical activity (Cardiac disorders) | 0 | 1
Right ventricular failure (Cardiac disorders) | 7 | 5
Supraventricular tachycardia (Cardiac disorders) | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Intussusception (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Rectal fissure (Gastrointestinal disorders) | 0 | 1
Adverse drug reaction (General disorders) | 0 | 1
Asthenia (General disorders) | 0 | 2
Chest pain (General disorders) | 2 | 2
Death (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 2 | 0
Impaired healing (General disorders) | 1 | 0
Infusion site reaction (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 3 | 1
Oedema peripheral (General disorders) | 1 | 1
Pyrexia (General disorders) | 2 | 0
Sudden cardiac death (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 1
Breast abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 3
Cellulitis (Infections and infestations) | 3 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1
Extradural abscess (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 0 | 5
Osteomyelitis (Infections and infestations) | 1 | 0
Osteomyelitis acute (Infections and infestations) | 1 | 0
Parotid abscess (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 8 | 12
Pneumonia influenzal (Infections and infestations) | 1 | 1
Pneumonia viral (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 1 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 2
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1
Adjacent segment degeneration (Injury, poisoning and procedural complications) | 1 | 0
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Shunt malfunction (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Anticoagulation drug level above therapeutic (Investigations) | 1 | 0
Electrocardiogram change (Investigations) | 0 | 1
Pulmonary arterial pressure increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 3 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Immunoglobulin G4 related disease (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Still's disease (Musculoskeletal and connective tissue disorders) | 0 | 1
Systemic scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 1
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vulval cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 4
Embolic cerebral infarction (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Post-traumatic epilepsy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 4 | 3
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 0 | 1
Generalised anxiety disorder (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 2 | 3
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
End stage renal disease (Renal and urinary disorders) | 1 | 0
Adenomyosis (Reproductive system and breast disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 23 | 30
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Aortic stenosis (Vascular disorders) | 1 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Esuberaprost (N=137) | Placebo (N=136)
Abdominal pain (Gastrointestinal disorders) | 10 | 7
Acute kidney injury (Renal and urinary disorders) | 5 | 7
Anaemia (Blood and lymphatic system disorders) | 12 | 8
Anxiety (Psychiatric disorders) | 3 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 12
Bronchitis (Infections and infestations) | 13 | 12
Cellulitis (Infections and infestations) | 10 | 3
Chest discomfort (General disorders) | 8 | 9
Chest pain (General disorders) | 5 | 7
Constipation (Gastrointestinal disorders) | 11 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 25
Decreased appetite (Metabolism and nutrition disorders) | 7 | 4
Depression (Psychiatric disorders) | 7 | 5
Diarrhoea (Gastrointestinal disorders) | 31 | 24
Dizziness (Nervous system disorders) | 24 | 36
Dyspepsia (Gastrointestinal disorders) | 6 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 35 | 42
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 9 | 6
Electrocardiogram QT prolonged (Investigations) | 7 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 8
Fall (Injury, poisoning and procedural complications) | 12 | 12
Fatigue (General disorders) | 22 | 28
Fluid overload (Metabolism and nutrition disorders) | 3 | 7
Flushing (Vascular disorders) | 17 | 17
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 | 3
Headache (Nervous system disorders) | 62 | 39
Hypokalaemia (Metabolism and nutrition disorders) | 14 | 7
Hypotension (Vascular disorders) | 4 | 9
Influenza (Infections and infestations) | 10 | 10
Insomnia (Psychiatric disorders) | 7 | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 11
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 14 | 12
Nasopharyngitis (Infections and infestations) | 20 | 19
Nausea (Gastrointestinal disorders) | 41 | 33
Non-cardiac chest pain (General disorders) | 8 | 8
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 18 | 10
Oedema (General disorders) | 6 | 9
Oedema peripheral (General disorders) | 22 | 17
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 7
Pain (General disorders) | 5 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 | 14
Pain in jaw (Musculoskeletal and connective tissue disorders) | 16 | 9
Palpitations (Cardiac disorders) | 14 | 14
Paraesthesia (Nervous system disorders) | 7 | 3
Pneumonia (Infections and infestations) | 11 | 6
Presyncope (Nervous system disorders) | 5 | 8
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 11 | 8
Pyrexia (General disorders) | 10 | 14
Respiratory tract infection (Infections and infestations) | 3 | 7
Sinusitis (Infections and infestations) | 21 | 19
Syncope (Nervous system disorders) | 9 | 8
Tooth infection (Infections and infestations) | 9 | 0
Upper respiratory tract infection (Infections and infestations) | 25 | 43
Urinary tract infection (Infections and infestations) | 25 | 20
Vomiting (Gastrointestinal disorders) | 15 | 16
Weight increased (Investigations) | 8 | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 7 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2014-10-15): https://cdn.clinicaltrials.gov/large-docs/99/NCT01908699/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-13): https://cdn.clinicaltrials.gov/large-docs/99/NCT01908699/SAP_001.pdf